CLINICAL TRIAL: NCT06031311
Title: Clinical Characteristics and Predictors of Pulmonary Hypertension in COPD at Different Levels of Smoking
Brief Title: Pulmonaryhypertension in Copd at Different Levels of Smoking
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrouk Mohamed Salah Mosleh, Resident doctor, Assiut University
Other Study IDs: Pulmonaryhypertension in copd
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography and HRCT — Echocardiography:is non invasive and easily accessible tool in the diagnosis of any patient with suspected PH.HRCT: is a non-invasive and easily accessible tool to detect pulmonary hypertension in COPD patients.

SUMMARY:
To identify Predictors of pulmonary hypertension in COPD patients and its relation to different levels of smoking

DETAILED DESCRIPTION:
COPD is a heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, expectoration and/or exacerbations) due to abnormalities of the airways (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow obstruction.It is also the most common cause of deaths in patients with chronic respiratory disease, the fatality rate in USA is 0.41%.Pulmonary Hypertension is the most common serious complication in COPD patients ; which occurs in up to 30% of patients and increases the mortality rate.Smoking is the leading cause of chronic obstructive pulmonary disease (COPD) Smoking is also a trigger for COPD flare-ups.Smoking damages the air sacs, airways, and the lining of your lungs. Injured lungs have trouble moving enough air in and out, so it's hard to breathe

ELIGIBILITY:
Inclusion Criteria:

* 1.All patients admitted to chest department or presented to our outpatient clinic with clinical and functional diagnosis of COPD among both sexes will be included 2.Age >18 years Old

Exclusion Criteria:

* 1.Patients under 18 years old. 2.pregnant patients. 3.patients with history hypertension or valvular diseases 4.Cardiomyopathic patient 5.Patients with concomitant obstructive sleep apnea 6.Patients with collagen vascular disease 7.Patients with thrombo-embolic disease 8. Patients with any chronic chest disease other than COPD

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Full clinical history including:[demographic data and clinical symptoms including cough with expectoration ,dyspnea,chest wheeze,…etc] 2.Full clinical examination. 3.laboratory investigations: Complete blood picture , kidney function test, liver function test,coagulation profile 4.Arterial blood gases [Pao2, Paco2,Sao2,Hco3, P(A_a)o2 ] 5.PFTS:will be performed and classified into: Post bronchodilator FEV1/FVC <0.7
  GOLD 1 - mild: FEV1 ≥80% predicted. GOLD 2 - moderate: 50% ≤ FEV1 <80% predicted. GOLD 3 - severe: 30% ≤ FEV1 <50% predicted. GOLD 4 - very severe: FEV1 <30% predicted [5] 6.Echocardiography:is non invasive and easily accessible tool in the diagnosis of any patient with suspected PH. ePASP is estimated by calculating Doppler estimated trans tricuspid gradient (TR gradient= 4 x (TR velocity)2) and adding estimated right atrial pressure to it based on the size of the inferior vena cava and collapsibility.[6]
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Predictors of pulmonary hypertension in COPD patients | 1 year
  Predict pulmonary hypertension in COPD patients

SECONDARY OUTCOMES:
Relationship between different levels of smoking and predictors of degree of pulmonary hypertension | 1 year
  Levels of smoking (mild.moderate.sever.non smoker) and it's relation to pulmonary hypertension in COPD patients

REFERENCES:
- See also: Global Initiative for Chronic Obstructive Lung Disease 2023 — https://goldcopd.org/2023-gold-report-2/